CLINICAL TRIAL: NCT04956809
Title: Effect of Dapagliflozin on Submaximal Exercise Tolerance in Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Kenneth B Margulies, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 848538
Record Dates: First submitted 2021-06-30; First posted 2021-07-09 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: HFrEF
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin 10mg (Active Comparator): Active arm will be 6 weeks in duration, separated by a 2-week wash-out period.
  Interventions: Drug: Dapagliflozin 10Mg Tab
- Placebo (Placebo Comparator): Placebo arm will be 6 weeks in duration, separated by a 2-week wash-out period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10Mg Tab — This will be a single-center randomized, placebo controlled, double-blind, 2-treatment, 2-phase cross-over trial in 27 HFrEF subjects: (A) Dapa 10 mg daily; (B) Placebo.
  Arms: Dapagliflozin 10mg
Drug: Placebo — This will be a single-center randomized, placebo controlled, double-blind, 2-treatment, 2-phase cross-over trial in 27 HFrEF subjects: (A) Dapa 10 mg daily; (B) Placebo.
  Arms: Placebo

SUMMARY:
This study will examine whether and how the FDA-approved drug dapagliflozin (Dapa) improves submaximal exercise endurance and skeletal muscle oxidative phosphorylation capacity (SkM OxPhos) in patients with heart failure and reduced left ventricular ejection fraction (HFrEF).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of HFrEF with NYHA Class II-III functional class, which has been present for at least two months
2. Left ventricular ejection fraction ≤ 40%
3. Stable medical therapy for at least 1 month
4. Plasma NT-proBNP level of: ≥ 200pg/mL; OR ≥ 125pg/mL if they were hospitalized for HF within the past 12 months; or ≥ 250 pg/mL if patient had atrial fibrillation/flutter on baseline ECG

Exclusion Criteria:

1. Receiving therapy with an SGLT2 inhibitor within 8 weeks prior to enrollment or previous intolerance of an SGLT2 inhibitor
2. Type 1 diabetes mellitus
3. Age <18 years old
4. Pregnancy: Women of childbearing potential will undergo a urine pregnancy test during the screening visit.
5. Uncontrolled atrial fibrillation, as defined by a resting heart rate > 100 beats per minute at the time of the baseline assessment
6. Paroxysmal atrial fibrillation (Afib) or flutter with >1 hour of continuous Afib documented within the previous 6 months (prior to screening or randomization), direct-current (DC) cardioversion or ablation procedure for Afib within 6 months, or plan to attempt to restore sinus rhythm (with drug therapy, ablation, or DC cardioversion) within 6 months of randomization. Subjects with persistent Afib and no sinus rhythm documented in the prior 6 months are permitted.
7. Hemoglobin < 10 g/dL
8. eGFR < 25 mL/min/1.73m^2, or unstable or rapidly progressing renal disease at the time of randomization
9. Subject inability/unwillingness to exercise
10. Greater than moderate left sided valvular disease (mitral regurgitation, aortic stenosis, aortic regurgitation), moderate or greater mitral stenosis, severe right-sided valvular disease
11. Known hypertrophic, infiltrative, restrictive or inflammatory cardiomyopathy
12. Clinically significant pericardial disease, as per investigator judgment
13. Current angina due to clinically significant epicardial coronary disease, as per investigator judgment
14. Acute coronary syndrome or coronary intervention within the past 2 months
15. Primary pulmonary artery hypertension (WHO Group 1 Pulmonary Arterial Hypertension)
16. Clinically significant lung disease as defined by: Chronic Obstructive Pulmonary Disease meeting Stage III or greater GOLD criteria (FEV1<50% predicted), treatment with oral steroids within the past 6 months for an exacerbation of obstructive lung disease, current use of supplemental oxygen aside from nocturnal oxygen for the treatment of obstructive sleep apnea.

    - Desaturation to <90% on the baseline maximal effort cardiopulmonary exercise test will also be grounds for exclusion
17. Clinically-significant ischemia, as per investigator's judgement, on stress testing without either (1) subsequent revascularization, (2) an angiogram demonstrating the absence of clinically significant epicardial coronary artery disease, as per investigator judgment; (3) a follow-up 'negative' stress test, particularly when using a more specific technique (i.e., a negative perfusion imaging test following a 'positive' ECG stress test)

    - Exercise induced regional wall motion abnormalities suggestive of ongoing ischemia during the baseline maximal effort cardiopulmonary exercise test will be exclusionary
18. Implantation of a CRT device within 12 weeks prior to enrollment or intent to implant a CRT device during the study period
19. Previous cardiac transplantation or implantation of a ventricular assist device, or implantation expected after randomization
20. Symptomatic bradycardia or second- or third-degree heart block, in the absence of a pacemaker
21. Significant liver disease impacting synthetic function or volume control (ALT/AST > 3x ULN, Albumin < 3.0 g/dL)
22. Severe right ventricular dysfunction
23. Baseline resting seated systolic blood pressure > 180 mmHg or <90 mmHg
24. Orthostatic blood pressure response to the transition from supine to standing (>20 mmHg reduction in systolic blood pressure 2-3 minutes after standing)
25. Active participation in another study that utilizes an investigational agent (observational studies/registries allowed)
26. Any condition that, in the opinion of the investigator, will interfere with the completion of the study. This may include comorbid or psychiatric conditions that may impede successful completion of the protocol, or logistical concerns (e.g. inability to travel to the exercise unit).

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the change in submaximal exercise endurance (time to exhaustion at 75% of peak workload) between Dapa and placebo. | 24 Months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No